CLINICAL TRIAL: NCT01840332
Title: Method of Endogenous TSH Stimulation in the Follow-up of Differentiated Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Vallo Volke, Dr., University of Tartu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1.0 /29.08.2012
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L-thyroxin (Experimental): this is one arm study
  Interventions: Drug: L-thyroxin

INTERVENTIONS:
Drug: L-thyroxin — Low dose of L-thyroxin (50 microg/day) will be used during 4 weeks. If TSH is < 30 after 4 weeks the study continues up to 6 weeks.

SUMMARY:
The treatment of differentiated thyroid cancer (DCT) includes surgery followed by radioiodine treatment. In the follow-up of patients it is necessary to induce TSH elevation to test for cancer recurrence. One of the options is to stop L-thyroxin replacement for several weeks. Current pilot study aims to induce the necessary TSH elevation by decreasing the L-thyroxin dose. The main hypothesis is that necessary TSH stimulation will be achieved during 4-6 weeks in majority of patients.

DETAILED DESCRIPTION:
The treatment of differentiated thyroid cancer (DCT) includes surgery followed by radioiodine treatment. In the follow-up of patients it is necessary to induce TSH elevation for the measurement of thyreoglobulin and/or total body scanning. There are two principal methods to obtain TSH elevation: 1) injection of recombinant human TSH , and 2) to stop L-thyroxin replacement for several (3-4) weeks. As use of recombinant TSH is rather expensive, this method is not feasible in many countries. The problem with stopping L-thyroxin is development of severe hypothyroidism for several weeks with concomitant symptoms and signs.

Current pilot study aims to induce the necessary TSH elevation by decreasing the L-thyroxin dose. The main hypothesis is that necessary TSH stimulation will be achieved during 4-6 weeks in majority of patients with fixed dose of L-thyroxin. Concomitantly, blood tests and symptoms and signs of hypothyroidism will be obtained to get information about possible deviations during treatment with low dose of thyroxin.

ELIGIBILITY:
Inclusion Criteria:

* Differentiated thyroid cancer
* treated by thyroidectomy and at least 1 ablation with 131-I > 5 months ago
* TSH < 4 imU/L

Exclusion Criteria:

* Pregnancy
* Known metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
TSH level at the end of study | 4-6 weeks
  The percentage of patients obtaining TSH level at least 30 imU/L at the end of study period.
  Blood tests will be obtained after 4 weeks. If TSH > 30 the patient has completed the study. If TSH < 30 patient will continue for 1 week and blood tests will be obtained after week 5. If TSH > 30 the patient has completed the study. If TSH < 30 patient will be monitored during 1 week and blood tests will be obtained after 6 weeks.

SECONDARY OUTCOMES:
change in Billewitz index during the study | 4-6 weeks
  Billewitz index measures the severity of hypothyroidism symptoms. Billewitz index will be recorded after 4 weeks and after 5 and 6 weeks if patient continues after 4 or 5 weeks (see primary endpoint for details).

OTHER OUTCOMES:
change in biochemical parameters during the study | 4-6 weeks
  Change in parameters related to hypothyroidism (thyroid hormones, creatinine kinase, cholesterol,ultra sensitive CRP, creatinine).

CONTACTS AND LOCATIONS:
Overall Officials: Vallo Volke, MD, PhD, Principal Investigator — University of Tartu
Locations (2):
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu